CLINICAL TRIAL: NCT00066911
Title: Functional Brain Mapping of Laryngeal Sensorimotor Control in Voice Disorders
Brief Title: Brain Mapping of Voice Control
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030260; 03-N-0260
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-11-05

CONDITIONS: Voice Disorders
Keywords: Functional Magnetic Resonance Imaging; Vocalization; Spasmodic Dysphonia; Muscular Tension Dysphonia; Topical Lidocaine; Voice Disorders; Vocal Tremor; Healthy Volunteer; HV
MeSH Terms: conditions — Voice Disorders; Dysphonia

SUMMARY:
Some voice disorders are caused by uncontrolled muscle actions that affect the larynx or voice box.

The purpose of this study is to understand 1) how the brain controls voice production; 2) how changes in sensation within the voice box affect brain control of the voice box; 3) how the central nervous system is affected when people have motor or sensory abnormalities that affect the voice box; and 4) whether patients with voice disorders differ from people without voice disorders in the way the brain controls the voice box. By better understanding these concepts, researchers hope to develop improved treatments for patients with voice disorders.

Forty-five healthy adult volunteers and 90 patients with voice disorders will participate in this study. Participants must be between the ages of 20 and 70. The study will involve two visits to the Clinical Center. During the first visit, participants will undergo a medical history and physical exam. During the second visit, investigators will perform the following procedures on study participants: 1) look at the voice box with a nasolaryngoscope, a fine tube through the nose; 2) use MRI [magnetic resonance imaging] to record brain activity while participants use their voice to speak; 3) changing sensation in the voice box by dripping a topical anesthetic onto the vocal folds; and 4) using MRI to again record brain activity during speech immediately after applying the topical anesthetic.

Participants will receive up to $700 in compensation for their involvement in this study.

DETAILED DESCRIPTION:
The neural organization of laryngeal motor and somatosensory function will be investigated in adults with idiopathic voice disorders using functional magnetic resonance imaging. Brain activation will be compared in normal volunteers and patients with spasmodic dysphonia (SD), muscle tension dysphonia (MTD) and vocal tremor. While each voice disorder is characterized by strained vocalization, the disorders are distinguished by other differences in voice symptoms. Accordingly, the brain correlates of vocalization in these disorders may both differ from each other and that of normal vocal function. Because sensory feedback has been identified as a factor in SD, the role of afferent input in vocalization will be investigated by comparing brain activation before and after topical anesthesia of the laryngeal mucosa. The afferent blockade is expected to significantly suppress dysphonic symptoms in SD patients for the duration of the block. The change in symptomatology may be associated with a temporary but significant change in central sensorimotor patterns in these patients. The block is not expected to alter MTD, vocal tremor or normal vocal function. The brain activation changes that accompany symptom relief in SD patients will determine alterations in central neural control that have a role in symptom generation in SD. Identifying these differences in central sensorimotor control between the disorders will provide insight into their differences in pathophysiology.

Objectives:

1. To determine if emotional vocalization and linguistic vocalization involve different cortical and sub-cortical functional networks in normal adults.
2. To determine if only the brain activation network active for linguistic vocalization network differs between normal controls and dysphonia patients during equivalent voice production effort.
3. To determine if patients with dysphonia differ from controls during the performance of non-vocal laryngeal gestures when patients are asymptomatic.
4. To determine if a reduction in sensation during topical anesthesia alters linguistic vocalization in dysphonia but not in controls.

ELIGIBILITY:
* INCLUSION CRITERIA:

The inclusion criteria for normal volunteers are normal vocal function and average health as determined by the staff otolaryngologist. Normal vocal function refers to normal voice quality, a negative history for voice or laryngeal disorders. Persons with significant pulmonary, neurological and psychiatric function will not be recruited. The primary inclusion criteria for the voice disordered groups are a current diagnosis of spasmodic dysphonia (abductor or adductor type), muscular tension dysphonia or voice tremor. These persons will not have pulmonary, neurological or psychiatric disorders or exclusion criteria.

INCLUSION CRITERIA - for Patients with Spasmodic Dysphonia:

Intermittent strained hoarseness, uncontrolled voice breaks or changes in pitch are present during vowels, liquids (r & l) and semi-vowels (w & y), during speech for adductor SD or prolonged voiceless consonants producing breathy breaks for abductor SD;

Less prominent symptoms during whisper, singing or falsetto,

Normal voice and vocal fold movement for protective and emotional laryngeal function, such as cough, laugh or cry;

A diagnosis of adductor or adductor spasmodic dysphonia based on voice testing and fiberoptic nasolaryngoscopy by a board certified otolaryngologist and Speech-Language Pathologist during the initial interview;

Exclusion of other laryngeal pathologies based on a fiberoptic nasolaryngoscopic examination conducted during the initial interview by the staff otolaryngologist.

INCLUSION CRITERIA - for Patients with Muscular Tension Dysphonia:

Increased phonatory muscle tension in the paralaryngeal and suprahyoid muscles on palpation;

A consistent hypertonic laryngeal posture for phonation, such as either an anterior-posterior squeeze (pin-hole posture) or ventricular hyper adduction and an absence of SD or vocal tremor as determined by a Speech-Language Pathologist and the staff otolaryngologist;

Exclusion of other laryngeal pathologies based on a fiberoptic nasolaryngoscopic examination conducted during the initial interview by the staff otolaryngologist.

INCLUSION CRITERIA - for Patients with Vocal Tremor:

Vocal tremor during vocalization that primarily involves laryngeal structures;

Exclusion of other laryngeal pathologies based on a fiberoptic nasolaryngoscopic examination conducted during the initial interview by the staff otolaryngologist.

EXCLUSION CRITERIA:

Any individual with a history of one or more of the following contraindications will be excluded from the study:

Airway obstruction, smoking or tobacco use;

Pulmonary, or neurological disease;

Pregnancy as reported by the volunteer or a positive pregnancy result from a urine sample obtained on the day of testing;

Psychiatric disorder, under psychiatric care, or on medication for psychiatric disorders. Examples of psychiatric disorders to be excluded are: somatoform disorders, conversion disorders, major depression, schizophrenia or a bipolar disorder. A history of a previous episode of minor reactive depression would not exclude a person from participation;

Speech or hearing problems as determined by medical history and examination by the otolaryngologist. A 30 dB HL hearing screening between 500 and 3000 Hz will be conducted if subjects report difficulty following spoken instructions or significant noise exposure;

A reduction in the range of vocal fold movement during non-speech tasks such as whistling suggesting either paralysis or paresis, joint abnormality or neoplasm as determined by videolaryngoscopic examination by the staff otolaryngologist;

Complete aphonia, a history of airway obstruction or structural abnormalities affect the larynx such as vocal fold nodules, polyps, carcinoma, cysts, contact ulcers, chronic laryngitis as determined by videolaryngoscopic examination by the staff otolaryngologist;

Individuals having any condition that would present unnecessary risk to them, e.g., claustrophobia.

Specific contraindications for magnetic resonance imaging include: i) Any implant or surgical clip - implanted neural stimulator, implanted cardiac pacemaker or autodefibrillator, cochlear implant, ocular implant, aneurysm clip, artificial heart valve, insulin pump, orthopedic pins or prosthesis; ii) Any ferromagnetic foreign body - metal shavings, shrapnel, orthodontic braces, certain tattoos or permanent eye liner; and, iii) Any other implanted device or foreign body not listed above that is possibly ferromagnetic.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174
Dates: Start 2003-08-02; Primary Completion 2009-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ludlow CL, Schulz GM, Yamashita T, Deleyiannis FW. Abnormalities in long latency responses to superior laryngeal nerve stimulation in adductor spasmodic dysphonia. Ann Otol Rhinol Laryngol. 1995 Dec;104(12):928-35. doi: 10.1177/000348949510401203. PMID 7492063
- [Background] Dworkin JP, Meleca RJ, Simpson ML, Garfield I. Use of topical lidocaine in the treatment of muscle tension dysphonia. J Voice. 2000 Dec;14(4):567-74. doi: 10.1016/s0892-1997(00)80012-0. PMID 11130113
- [Background] Jurgens U. Neural pathways underlying vocal control. Neurosci Biobehav Rev. 2002 Mar;26(2):235-58. doi: 10.1016/s0149-7634(01)00068-9. PMID 11856561